CLINICAL TRIAL: NCT02533336
Title: The Effectiveness of Non-Pyrethroid Insecticide-Treated Durable Wall Liners as a Method for Malaria Control in Endemic Rural Tanzania: Cluster Randomized Trial
Brief Title: The Effectiveness of Non-Pyrethroid Insecticide-Treated Durable Wall Liners as a Method for Malaria Control in Endemic Rural Tanzania
Acronym: DL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: futility ground
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); London School of Hygiene and Tropical Medicine (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Brandeis University (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Geofrey Makenga, Research Scientist, National Institute for Medical Research, Tanzania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DL Project in Tanzania
Record Dates: First submitted 2014-07-13; First posted 2015-08-26 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Malaria
Keywords: Malaria control; Insecticide treated durable Wall Liners; Malaria incidence; Randomized Trial
MeSH Terms: conditions — Malaria | interventions — abamectin; fenpyroximate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DL+LLINs (Experimental): DL treated with abamectin and fenpyroximate
  Interventions: Drug: abamectin and fenpyroximate
- LLINs (No Intervention): LLINs only

INTERVENTIONS:
Drug: abamectin and fenpyroximate
  Arms: DL+LLINs

SUMMARY:
Over one year period in an area with universal coverage of LLIN and ACT provision as the first-line treatment of malaria, the investigators intend to evaluate the impact of DL on malaria transmission as measured by the incidence of malaria parasitemia, the prevalence of moderate to severe anemia, and entomological parameters. Information on the relative cost-effectiveness estimates of DL and the community acceptability of DL will also be measured.

DETAILED DESCRIPTION:
Vector control, together with prompt treatment with an artemisinin-based combination therapy (ACT) for individuals diagnosed with malaria and intermittent preventive treatment in pregnant women, is a critical component of malaria control in Africa. The two main vector control interventions used in Africa are long-lasting insecticidal nets (LLINs) and indoor residual spraying (IRS). LLINs are currently the mainstay of vector control and are believed to have contributed to the recent dramatic decline in malaria cases. However, resistance to the pyrethroid insecticides used in the bed nets has increased. The second main vector control method, IRS, has been an extremely effective adjunct to LLINs; its usefulness is threatened by the high cost of repeated applications and increasing mosquito resistance to insecticides used for spraying.

A new product, durable lining (DL) treated with non-pyrethroid insecticides, has been developed by Vestergaard, which theoretically mimics the effect of IRS but is designed to last for a minimum of three years. The product consists of a mixture of two non-pyrethroid insecticides incorporated into a polymer fabric that are designed to migrate differentially over the lifetime of the product to ensure sustained bioefficacy. The use of two agents may also decrease the risk of development of resistance. It is estimated that the cost of the insecticide treated wall liners (DL), which are installed on the indoor walls of houses, would be equal to 2-3 rounds of IRS.

To test the effectiveness of this new product, we will conduct a two-arm controlled randomized cluster trial to test the hypothesis that DL + LLINs are superior to LLINs alone. Over twelve (12) months (August 2015- Aug 2016), in an area with universal coverage (UC) of LLINs and where artemisinin combination therapies (ACT) are provided as the first-line treatment of malaria, we intend to evaluate the impact of DL on malaria transmission among children ages 6 months to 11 years as measured by the incidence of malaria parasitemia (symptomatic and asymptomatic), and the prevalence of moderate to severe anemia in under-fives. In addition, we will assess the effect of DL on entomological parameters, and measure the acceptability and a cost-effectiveness of the intervention. Stratified randomization based on malaria prevalence during the baseline survey will be used to select 22 clusters per arm in Muheza district.

ELIGIBILITY:
Inclusion criteria:

* Permanent residence in a selected household
* Aged 6 months- 11years for cohort study
* Informed parental consent
* For children between 8-11 years old, written assent

Exclusion criteria:

* Severely ill and unlikely to be able to complete the study
* Family does not intend to remain in the study area during the study period, or through the long rains
* Household does not accept intervention
* Not living in the study area when interventions were implemented
* enrolled in other interventional study

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4917 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of malaria parasitemia | 1 year
  The primary end point of the study is the cumulative incidence of malaria parasitaemia (asymptomatic or symptomatic) defined as the number of mRDT-confirmed episodes of parasitaemia per person-year

SECONDARY OUTCOMES:
Effectiveness of DL on anemia | 1 year
  change in mean haemoglobin in the intervention arm compared to the control

CONTACTS AND LOCATIONS:
Overall Officials: William N Kisinza, PhD, Principal Investigator — National Institute for Medical Research; Joseph P Mugasa, PhD, Study Director — National Institute for Medical Research
Locations (1):
- Muheza, Tanga, Muheza, Tanzania

REFERENCES:
- [Derived] Mpangala KR, Halasa-Rappel YA, Mohamed MS, Mnzava RC, Mkuza KJ, Mangesho PE, Kisinza WN, Mugasa JP, Messenger LA, Mtove G, Kihombo AR, Shepard DS. On the cost-effectiveness of insecticide-treated wall liner and indoor residual spraying as additions to insecticide treated bed nets to prevent malaria: findings from cluster randomized trials in Tanzania. BMC Public Health. 2021 Sep 14;21(1):1666. doi: 10.1186/s12889-021-11671-2. PMID 34521374
- [Derived] Mtove G, Mugasa JP, Messenger LA, Malima RC, Mangesho P, Magogo F, Plucinski M, Hashimu R, Matowo J, Shepard D, Batengana B, Cook J, Emidi B, Halasa Y, Kaaya R, Kihombo A, Lindblade KA, Makenga G, Mpangala R, Mwambuli A, Mzava R, Mziray A, Olang G, Oxborough RM, Seif M, Sambu E, Samuels A, Sudi W, Thomas J, Weston S, Alilio M, Binkin N, Gimnig J, Kleinschmidt I, McElroy P, Moulton LH, Norris L, Ruebush T, Venkatesan M, Rowland M, Mosha FW, Kisinza WN. The effectiveness of non-pyrethroid insecticide-treated durable wall lining to control malaria in rural Tanzania: study protocol for a two-armed cluster randomized trial. BMC Public Health. 2016 Jul 25;16:633. doi: 10.1186/s12889-016-3287-3. PMID 27456339